CLINICAL TRIAL: NCT00778752
Title: Dose-finding Study of Lenalidomide as Maintenance Therapy in Multiple Myeloma After Allogeneic Stem Cell Transplantation
Brief Title: Dose-finding of Lenalidomide as Maintenance in Multiple Myeloma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Revlimid as maintenance in MM
Record Dates: First submitted 2008-10-22; First posted 2008-10-23 (Estimated); Last update posted 2015-05-13 (Estimated); Status verified 2015-05

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Stem Cell Transplantation; Revlimid; Lenalidomide
MeSH Terms: conditions — Multiple Myeloma | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): Lenalidomide-treatment starts between 100 and 180 days after allogeneic stem cell transplantation. Three dose-levels will be investigated.
  * Dose-level -1: 2.5 mg/d if 2.5mg capsules are available, day 1-21, otherwise 5 mg every other day, day 1-21
  * Dose-level 0: 5 mg/d, day 1-21
  * Dose-level 1: 10 mg/d, day 1-21
  * Dose-level 2: 15 mg/d, day 1-21
  Interventions: Drug: Revlimid (Lenalidomide)

INTERVENTIONS:
Drug: Revlimid (Lenalidomide) — 3 pat. will be enrolled on dose level 0. If no DLTs are observed during cycles 1+2 dose will be escalated to the next higher level in the 3 patients. If 1 of 3 pat. experiences DLT at the current dose, then up to 3 more pat. will be accrued at the same level. If none of these 3 additional pat. experience DLT dose will be escalated in subsequent patients. If 1 of these 3 patients experiences DLT, the next lower level will be declared to be MTD and the study will be filled up with patients at this dose level up to 25 pat. overall.
  If 2 or more of 3 pat. or 3 or more of 6 pat. in the same cohort encounter DLT, the MTD has been exceeded and the previous lower dose level will be declared as MTD and the study will be filled up with patients at this level up to 25 pat. overall.
  If DLT is observed in level 0, the next dose level will be -1 for the following cohort of 3 patients. If level 2 is well tolerated without DLT, this level will be claimed as recommended dose for further trials.

SUMMARY:
This study is a Phase I (non-randomized) study evaluating three dose-levels of Lenalidomide in patients after allogeneic stem cell transplantation, accomplished in two institutions (University Medical Center Hamburg-Eppendorf/ University Medical Center Heidelberg).

ELIGIBILITY:
Inclusion Criteria:

* Understand and voluntarily sign informed consent form
* Age > 18 years at the time of signing the informed consent form
* Able to adhere to the study visit schedule and other protocol requirements
* Multiple myeloma patients who received allogeneic stem cell transplantation (100 to 180 days ago)
* No active acute GvHD (grade II - IV)
* No active infectious complications
* ECOG performance status of < 2 at study entry
* Laboratory test results within these ranges:

  * Absolute WBC count > 3.0 x 10^9/l
  * Platelet count > 80 x 10^9/l
  * Serum creatinine < 1.5 mg/dl
  * Total bilirubin < 1,5 mg/dl
  * AST (SGOT) and ALT (SGPT) < 3 x ULN
* Females of childbearing potential must agree to use two reliable forms of contraception simultaneously or to practice complete abstinence from heterosexual intercourse for at least 28 days before starting study drug, while participating in the study and at least 28 days after discontinuation from the study.
* male subjects must agree to use a latex condom during sexual contact with females of childbearing potential while participating in the study and for at least 28 days after discontinuation of study drug
* disease free of prior malignancies for > 5 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "in situ" of the cervix or breast

Exclusion Criteria:

* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form
* pregnant or breast feeding females
* use of any other experimental drug or therapy within 28 days of baseline
* known hypersensitivity to thalidomide
* concurrent use of other anti-cancer agents or treatments
* known positive for HIV of infectious hepatitis, type A, B, or C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-04; Primary Completion 2013-03 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Maximal tolerable dose of lenalidomide after allogeneic stem cell transplantation in patients with multiple myeloma | 2 years post-transplantation

SECONDARY OUTCOMES:
Determination of remission status after lenalidomide treatment | 2 years post-transplantation
Effect on T-cell/ NK-cell recovery | 1 year post-transplantation
Incidence of infectious complications and GvHD | 1 year post-transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Nicolaus Kroeger, Prof. Dr., Principal Investigator — University Medical Center Hamburg-Eppendorf, Germany
Locations (2):
- Germany (2):
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Universitätsklinikum Heidelberg, Heidelberg

REFERENCES:
- [Derived] Wolschke C, Stubig T, Hegenbart U, Schonland S, Heinzelmann M, Hildebrandt Y, Ayuk F, Atanackovic D, Dreger P, Zander A, Kroger N. Postallograft lenalidomide induces strong NK cell-mediated antimyeloma activity and risk for T cell-mediated GvHD: Results from a phase I/II dose-finding study. Exp Hematol. 2013 Feb;41(2):134-142.e3. doi: 10.1016/j.exphem.2012.10.004. Epub 2012 Oct 17. PMID 23085463